CLINICAL TRIAL: NCT04046536
Title: rTMS in Alleviating Pain and Co-morbid Symptoms in GWVI
Brief Title: rTMS in Alleviating Pain and Co-Morbid Symptoms in Gulf War Veterans Illness (GWVI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPLD-013-18F; H190020 (Other: VASDHS)
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Gulf War Illness; Depression
Keywords: rTMS; Transcranial Magnetic Stimulation; Gulf War Illness; Depression
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: There will be two groups: one will receive active rTMS and the other group will receive sham rTMS.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blinded study where only the statistician is aware of the randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Active rTMS at the LDLPFC (Active Comparator): Subjects will receive the repetitive Transcranial Magnetic Stimulation (rTMS) study procedure at the left dorsolateral prefrontal cortex (LDLPFC).
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham rTMS at the LDLPFC (Sham Comparator): Sham rTMS will appear the same as the active, with the same parameters, but will not receive the actual magnetic stimulation to the LDLPFC.
  Interventions: Device: Sham Transcranial Magnetic Stimulation
- Active rTMS at the LMC (Experimental): Subjects will receive the repetitive Transcranial Magnetic Stimulation (rTMS) study procedure at the left motor cortex (LMC)
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham rTMS at the LMC (Experimental): Sham rTMS will appear the same as the active, with the same parameters, but will not receive the actual magnetic stimulation to the LMC.
  Interventions: Device: Sham Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — A non-invasive treatment that emits magnetic pulses to stimulate the brain.
  Arms: Active rTMS at the LDLPFC; Active rTMS at the LMC
Device: Sham Transcranial Magnetic Stimulation — Sham rTMS will consist of the same parameters as active, however, the subject will not receive the actual magnetic stimulation due to the use of a double sided Active/Sham coil used specifically for research studies.
  Arms: Sham rTMS at the LDLPFC; Sham rTMS at the LMC

SUMMARY:
This study aims to look at the effectiveness of using repetitive transcranial magnetic stimulation (rTMS) in relieving pain and other co-morbid symptoms of Gulf War Illness.

DETAILED DESCRIPTION:
Headaches (HA), muscle and joint pain, are some of the most common debilitating symptoms in military personnel served in the 1990-1991 Persian Gulf War (GW1). Migraine like HA and diffuse body pain were detected in 64% of Gulf War Veteran (GWV) diagnosed with Gulf War Illness (GWI). Likewise, depression carries a very high co-morbid rate (50%) in patients with chronic pain, and in GWV with GWI related chronic HA and body muscle and joint pain conditions (GWI-HAP). Unfortunately, conventional pharmacological treatments for GWI-related pain has not been shown to be effective and drugs such as narcotics contain many long term untoward psychosomatic and abusive side effects. This study is assessing the effectiveness of repetitive transcranial magnetic stimulation (rTMS), non-invasive treatment option, in alleviating pain and other co-morbid symptoms of GWI.

ELIGIBILITY:
Inclusion Criteria:

* Male or female under 65 years of age who served in the military for at least 30 consecutive days between August 1, 1990, and July 31, 1991 in the Persian Gulf War region
* CDC Criteria for GWVI (GWI)
* Kansas Criteria for GWVI (GWI)
* International Headache Society Criteria for Migraine Headache without aura
* Average Overall Daily Muscle Pain Intensity >3 on 0-10 a NPS
* Average Overall Daily Extremities Joint Pain Intensity >3 on 0-10 a NPS
* Headache Exacerbation/attack once a week with the average intensity >3 on a 0-10 NPS, lasting > 1 hour in the past three months
* Hamilton Rating Scale of Depression (HRSD) greater than or equal to 14 based on the sum of scores for the first 17 items

Exclusion Criteria:

* Pregnancy
* History of pacemaker implant
* Any ferromagnetic (e.g. bullet fragment, shrapnel, device implant) in the brain or body that will prohibit the patients from having a brain MRI
* History of dementia, major psychiatric diseases, or life-threatening diseases
* Presence of any other chronic neuropathic pain states such as Complex Regional Pain Syndrome or Painful Peripheral Neuropathy
* History of seizure
* Pending litigation
* Low back pain with mechanical origins such as lumbar radiculopathy or radiculitis or lumbar facet arthropathy
* Lack of ability to understand the experimental protocol and to adequately communicate in English
* History of Traumatic Brain injury
* Chronic Tension or Cluster Headache
* Ongoing Cognitive Rehabilitation or Treatment of PTSD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to post treatment of GWI-related pain and headaches | Baseline, 1-week, 1-month, 2-month, and 3-month
  This outcome will be measured through daily self-reporting logs that tracks headache, muscle, and joint pain. A numerical rating scale of 0, being no pain, to 10, being worst possible pain, will be used to report pain and headaches.
Change from baseline to post treatment of sensory and affective aspects of pain | Baseline, 1-week, 1-month, 2-month, and 3-month
  Short Form McGill Pain Questionnaire (SF-MPQ): This is a self-report questionnaire that allows individuals to describe the quality and intensity of pain they are experiencing. This will be used to assess the sensory and affective aspects of muscle and joint pain.
Change from baseline to post treatment of headaches | Baseline, 1-week, 1-month, 2-month, and 3-month
  The Headache Impact Test (HIT-6) will be used to measure how headaches affect the individual's ability to function in different domains. This 6-question form assesses the severity of headache pain and is scored with a range of 36-78, with higher scores indicating a larger impact of headaches on functionality.
Change from baseline to post treatment of depression | Baseline, 1-week, 1-month, 2-month, and 3-month
  The Hamilton Rating Scale for Depression (HRSD) questionnaire will be used to assess depression, which consists of 21 questions and rates the severity of symptoms observed in depression such as low mood, insomnia, agitation, anxiety and weight loss. Only the first 17 items are used for the overall scoring. A score between 14 and 18 represents a moderate form of depression and a score greater than 19 represents severe depression.
Change from baseline to post treatment of quality of life | Baseline, 1-week, 1-month, 2-month, and 3-month
  The Short Form Health Survey-36 (SF-36) is a self-reported survey of patient health. It is a measure of health status and quality of life in regards to eight main areas: vitality, physical functioning, bodily pain, health perceptions, physical, emotional, and social role functioning and mental health.
Change from baseline to post treatment of body pain | Baseline, 1-week, 1-month, 2-month, and 3-month
  A Brief Pain Inventory-Short Form (BPI-SF) questionnaire will also be used to assess the severity of pain and the impact of pain on daily functions. The BPI-SF consists of five questions. Four items measure pain on 11-point response scales from 0 to 10 ("No Pain" to "Pain as bad as you can imagine". Another item, containing 7 sub-questions, evaluates the level of pain interference with daily functioning on 11-point response scales from 0 to 10 ("Does not interfere" to "Completely interferes").
Change from baseline to post treatment of muscle pain | Baseline, 1-week, 1-month, 2-month, and 3-month
  The New Clinical Fibromyalgia Diagnostic Criteria - Part 1 will be used to assess muscle pain. Patients will be asked to rate the average (over the past 24 hours) intensity of muscle pain for up to 12 locations of the body.
Change from baseline to post treatment of fibromyalgia | Baseline, 1-week, 1-month, 2-month, and 3-month
  A Revised Fibromyalgia Impact Questionnaire will be used to evaluate the function, overall impact and symptoms of Fibromyalgia. There are a total of 21 questions, each with a range of 0-10, with 10 being either "very difficult" or "always."
Change from baseline to post treatment of neurobehavioral symptoms | Baseline, 1-week, 1-month, 2-month, and 3-month
  The Neurobehavioral Symptoms Inventory (NSI) is a self-report questionnaire on the severity of various behavioral symptoms and is measured using a 5-item scale. It asks the subjects to indicate the extent to which each symptom has disturbed them.
Change from baseline to post treatment of sleep quality | Baseline, 1-week, 1-month, 2-month, and 3-month
  The Pittsburgh Sleep Quality Index (PSQI) questionnaire has nineteen individual items which are used to generate seven composite scores on: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Questions are either free-response or have a range from 0-3, with 3 being "more frequent" or "very bad."
Change from baseline to post treatment of sleep difficulties | Baseline, 1-week, 1-month, 2-month, and 3-month
  The Insomnia Severity Index measures the severity of an individual's sleep difficulties. All questions range from 0-4 and the sum of the answers would give the total score. The total score range from 0-28.
Change from baseline to post treatment of fatigue | Baseline, 1-week, 1-month, 2-month, and 3-month
  The Flinders Fatigue Scale measures daytime fatigue associated with insomnia through a 7-item questionnaire. The questions range from 1-5, with 5 being "extremely" or "entirely."

SECONDARY OUTCOMES:
Change from baseline to post treatment of PTSD symptoms | Baseline, 1-week, 1-month, 2-month, and 3-month
  The Clinician-Administered PTSD Scale (CAPS-5), 30-item structured interview that can be used to diagnose PTSD and associated symptoms, will be used to assess PTSD symptoms
Change in opioid-based pain medication usage | Baseline, 1-week, 1-month, 2-month, and 3-month
  Medication assessment consists of daily chronic and breakthrough opioid usage for pain or headache. Average daily dosage will be converted to equal-potent oral Morphine Sulfate dosage based on the clinical opioid conversion table used by the VASDHS Pain Service and University of California, San Diego, Center for Pain Medicine. The study participants will be asked to remain on the same analgesic medication(s) during the study period but are allowed to titrate down their narcotic usage.
Explore changes in supraspinal resting state functional connectivity | Baseline and 1-week post treatment
  The outcome measure will be assessed through functional magnetic imaging scans and subsequent processing.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Yick Leung, MD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (3):
- United States (3):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT04046536/ICF_000.pdf